CLINICAL TRIAL: NCT05866237
Title: COVER-ME: Covid-19 Vaccination Coverage Among Underserved Populations: Developing and Evaluating Community-based Interventions in East London Minority Ethnicity (ME) Populations; Underserved Migrants and Persons With Low Income.
Brief Title: COVID-19 Vaccine Uptake Amongst Underserved Populations in East London
Acronym: COVER-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Social Action for Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 151164
Record Dates: First submitted 2023-05-05; First posted 2023-05-19 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; Influenza; Vaccination Refusal
Keywords: Vaccination
MeSH Terms: conditions — COVID-19; Influenza, Human; Vaccination Refusal

STUDY DESIGN:
Intervention Model Description: Clustered randomised control trial (as participants will be recruited from 6 GP practices)
Who Masked: Participant
Masking Description: Eligible patients to be randomised 1:1. None of these patients would have received the vaccine prior to entry to the study. These patients who are eligible for the intervention, randomised are to receive one of two workflows on an individual basis (standard of care or the PET).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individuals allocated to this group will be receiving care from their GP as well as the patient engagement tool (intervention). This will include messages being sent to patients in regards to vaccine information and uptake at different time points (three times).
  Interventions: Device: Patient Engagement tool
- Control Group (No Intervention): The individuals in this group will receive standard care from their GP and nothing additional to this.

INTERVENTIONS:
Device: Patient Engagement tool — The study intervention (PET) aims to increase uptake of vaccines that are already recommended through national guidance.The PET will help educate and inform individuals about the benefits of COVID-19 and Flu vaccinations through culturally adapted educational support, including content, design, mode and timing of delivery of messages (text, video or voice messages).
  Arms: Intervention group

SUMMARY:
This is a randomised controlled pilot study evaluating and assessing the feasibility of a co-designed PET. The PET was co-designed in the qualitative work packages with members of the community as well as healthcare professionals (Ethical approval: REF QMERC22.266) that precedes this pilot trial.

Eligible patients from six GP practises from Tower Hamlets and Newham will be randomised to the intervention or control during the study.

DETAILED DESCRIPTION:
It is imperative that local residents' views are heard, particularly in underserved communities, when trying to address poor vaccine uptake. We are interested to elicit a wide range of views, and channel these to co-design a feasible and acceptable intervention with community groups.

This intervention will be evaluated in this randomised pilot study to assess feasibility, practicality and acceptability. This will be in preparation of a fully powered randomised controlled trial to evaluate the efficacy afterwards.

Eligible patients at all n=6 practices will be enrolled into the study at two time points (see below). Patients will be individually randomised 1:1 to receive the PET or routine care. We will use the Appt-Health workflow tool for both groups, although patients in the control group will be monitored but will not receive additional interventions than routine care. The comparison between those randomised to the intervention or control group is envisaged to be the primary comparison in a subsequent trial to evaluate efficacy (vaccination uptake). Individual randomisation will be stratified by GP, using a random block allocation list implemented into the software used for the study.

Participating centres All practices will be selected based on list size (larger practices with >10,000 patients), technological and practice infrastructure and procedures (to ensure smooth operability of the PET), demography of the practice population (to ensure good representation of underserved population groups) and capability and capacity (decided by the practice and network leads).

Randomisation The practices will be randomised by the study statistician. Individuals will be randomised, stratified by centre, using randomised block randomisation list allocations in the practice software. This will be done on the same day or shortly after the eligible list is determined. The randomised allocation will be visible to staff, but we will use the feasibility study to explore ways of blinding staff and patients for the definitive study.

Data collection and Analysis Eligible patients will be identified through the practice IT system (EMISWeb). We will provide some initial support and training to enable practices to complete missing ethnicity data. However, patients with unknown ethnicity resident in areas with index of multiple deprivation greater than the bottom quintile would not be included. The database associated with the software will record randomisation group, and record of the intervention to each participant, as well as engagement with different aspects of the tool (see secondary outcomes).

For analysis, we will extract pseudo-anonymised data and storage in the CASTOR database and analyse this on a secure research database and environment within the Barts Cancer Centre network at QMUL. Ethics and information governance approval will be sought for this.

ELIGIBILITY:
Inclusion Criteria:

* • Patient registered at study site (included GP surgery)

  * Adult (aged 18y+) at time of randomisation
  * Eligible for COVID-19 and/or Flu vaccination (ie. Not received either a first, second or booster vaccination)

AND

From an underserved population group, defined

1. non-white ethnicity OR
2. resident in a postcode in the bottom 20% of index of multiple deprivation OR
3. Those receiving little or no income

We will determine age, ethnicity, post-code and immunisation status from the patients' EMIS records.

Exclusion Criteria:

* They are unable or unwilling to consent (including those who do not consent to text messaging; those who opt out from taking part in research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5903 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is vaccination uptake in patients individually randomised. | Through study completion, until 6 months follow-up (>180 days since randomisation).
  This will be measured as the number (percent) of relevant SNOMED codes in eligible patients. Uptake will be measured from the time that the eligible group in each practice is identified (and randomised) until 6 months follow-up (>180 days since randomisation).

SECONDARY OUTCOMES:
Acceptability of the intervention | at 6 months
  a. To patients: Proportion of patients randomised to the intervention who engage with the PET and / or linked patient resources, as determined by user statistics logged on the software for i. The SMS messaging tool (number of SMS sent) ii. Number (percent) of patients who view the linked patient awareness resources iii. Usage of the patient work list tool b. To staff: Number and proportion of eligible patients randomised to the intervention processed using the patient work list tool
Feasibility of the intervention and randomisation | 6 months
  1. Number and proportion of eligible patients randomised
  2. Clinical capacity: number of slots available for vaccination bookings for each GP surgery and each day, by appointment time
Feasibility of the study design for a subsequent trial | 6 months
  1. Number and proportion of patients with all inclusion / exclusion data available on the electronic health records
  2. Number and proportion of patients eligible for the intervention
  3. Number and proportion of patients randomised who are sent material from the intervention (letter / sms)
  4. Number and proportion of patients eligible by vaccination status (none, first, second, with booster or without booster)
  5. Number and proportion of patients who opt out for their data to be used or withdraw from the study
  6. Number and proportion of patients who consent for further questionnaires
  7. Number and proportion of patients who are booked for a vaccination appointment
  8. Number and proportion of patients who are categorised a "failed encounter" (not booked, no more action taken)

OTHER OUTCOMES:
Vaccination uptake in patients after 3- and 9-months follow-up (>90 and >270 days). This will be measured as the number (percent) of relevant SNOMED codes in eligible patients identified during the period. | Through study completion, after 3- and 9-months follow-up (>90 and >270 days)
  This will be measured as the number (percent) of relevant SNOMED codes in eligible patients identified during the period.
Mean vaccination rate after 3-, 6- and 9-months follow-up. | After 3-, 6- and 9-months follow-up
  his will be measured as the number of patients vaccinated divided by the follow-up time. Time is defined as time from randomisation until the earliest of vaccination, leaving the GP, withdraw

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Church Road Health, London
  - Glen Road Surgery, London
  - St Andrews Health Centre/ St Pauls Way Health Centre, London
  - St Stephen's Health Centre, London
  - Stratford Village Health Centre, London

IPD SHARING:
Plan to Share IPD: No
Data collected will anonymised and only available to people who are from the internal research team, and external collaborators mentioned. Anonymised data may be shared later on during dissemination through publications and conferences.

REFERENCES:
- [Derived] Chaudhry T, Tum P, Tam HZ, Brentnall A, Smethurst H, Kielmann K, Kunst H, Hargreaves S, Campbell CNJ, Griffiths C, Zenner D. COVER-ME: developing and evaluating community-based interventions to promote vaccine uptake for COVID-19 and influenza in East London minority ethnicity (ME) and underserved individuals - protocol for a pilot randomised controlled trial. BMJ Open. 2025 Mar 18;15(3):e092568. doi: 10.1136/bmjopen-2024-092568. PMID 40107676

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT05866237/SAP_000.pdf